CLINICAL TRIAL: NCT00613132
Title: Phase I Dose Escalation of Gleevec in Combination With RAD001 Plus Hydroxyurea for Patients With Recurrent Malignant Glioma
Brief Title: Ph I Gleevec in Combo w RAD001 + Hydroxyurea for Pts w Recurrent MG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annick Desjardins (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005875; 7020-07-32 (Other: Legacy ID)
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; GBM; Brain tumor; RAD0001; Hydroxyurea; Gleevec; Imatinib; Droxia; Everolimus; Hydrea; Hydroxycarbamide; Recurrent GBM; Imatinib mesylate; Glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Imatinib Mesylate; Everolimus; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pts receiving EIACDs
  Interventions: Drug: Gleevec, RAD001, and Hydroxyurea
- 2 (Experimental): Pts not receiving EIACDs
  Interventions: Drug: Gleevec, RAD001, and Hydroxyurea

INTERVENTIONS:
Drug: Gleevec, RAD001, and Hydroxyurea — Dose of Gleevec will be 400 mg in 1st cohort & will be increased to 600 mg po/day & then to 400 mg bid in successive cohorts. Prescribed dose should be administered orally, w large glass of water. Pts should not eat large or high fat meal within 1 hour before or after gleevec dosing. Doses of 600 mg or less should be administered once daily, whereas doses greater than 600 mg should be administered as equal doses twice day. It is recommended that pts take their prescribed Gleevec at same time that they take their prescribed RAD001 & hydroxyurea, however, 30-60 minute interval between agents is acceptable if required for practical or other compliance issues.
  Other Names: Gleevec-Imatinib-Imatinib mesylate; RAD001-Everolimus; Hydroxyurea-Droxia-Hydrea-Hydroxycarbamide

SUMMARY:
Primary objective To determine maximum tolerated dose & dose limiting toxicity of imatinib mesylate & RAD001 when combined w fixed doses of hydroxyurea among pts w recurrent GBM who are on & not on enzyme-inducing anti-convulsants including pts not on anti-epileptic drugs Secondary objective To assess safety & tolerability of imatinib mesylate in combo w RAD001 & hydroxyurea in this population To characterize single-dose & repeated-dose pharmacokinetic profiles of imatinib mesylate & RAD001 combo therapy in this pt population.

To assess antiangiogenic effects, pre- and post-treatment, of imatinib mesylate, RAD001 & hydroxyurea combo therapy, using DCE-MRI to evaluate changes in extent of vascular permeability, perfusion & relative tumor blood volume; to explore assessment of tumor cellularity & tumor cell death by changes in DWI-MRI as quantitated by apparent diffusion coefficient maps.

DETAILED DESCRIPTION:
This is open-label, single center, 1-arm ph I dose-escalation study of continuous, daily doses of imatinib mesylate & RAD001 administered orally in combination w fixed doses of hydroxyurea in adult pts w recurrent or relapsing glioblastoma multiforme. Study format includes classical "3+3" dose escalation design to determine MTD & DLT of imatinib mesylate + RAD001 when combined w hydroxyurea among GBM pts. Pts will be stratified based on whether they who are receiving EIACD & each stratum will independently dose escalate. Additionally, study will characterize safety, tolerability, biologic activity, & pharmacokinetic profile of this combo therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pts w confirmed GBM, GS, AA, AO & AOA are presenting in 1st, 2nd/3rd recurrence/relapse
* Pts without tumor biopsy <1 wk/surgical resection <2 wks prior to starting study drug
* For stratum of non-EIAED pts, each pts off all enzyme inducing anticonvulsants for >2 wks prior to starting study drug
* Pts should be on non-increasing dose of steroids for >7 days prior to obtaining baseline Gd-MRI of brain
* Pts should be on non-increasing dose of steroids for >7 days prior to starting study drug
* Pts w previous implantation of Gliadel may be eligible after discussion between investigator & sponsor
* Multifocal disease is eligible
* Age >18 yrs
* KPS >70
* Hematology: ANC>1.5 x 10^9/L, Hgb>9 g/dL, Platelets>100 x 10^9/L
* Biochemistry: K≥ LLN/correctable w supplement, Total Ca≥ LLN/correctable w supplement, Mg≥ LLN/correctable w supplement, P≥ LLN/correctable w supplement, AST/SGOT & ALT/SGPT <2.5 x ULN, Serum bilirubin <1.5 x ULN, Serum creatinine <1.5 x ULN/measured 24hr CrCl<0 mL/min/1.73m2, & Cholesterol≤ 00 mg/dL & triglyceride≤2.5 ULN
* Life expectancy ≥12wks
* Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

* Pts w any peripheral neuropathy ≥CTCAE gr2
* Pts w unresolved diarrhea ≥CTCAE gr2
* History of impaired cardiac function
* Obligate use of cardiac pacemaker, Congenital long QT syndrome, History or presence of ventricular or atrial tachyarrhythmias, Clinically significant resting bradycardia , Right bundle branch block + left anterior hemiblock
* Other clinically significant cardiac diseases
* Uncontrolled Db
* Active or uncontrolled infection requiring intravenous antibiotics
* Impairment of GI function/GI disease that may significantly alter absorption of Gleevec, hydroxyurea and/or RAD001
* Acute/chronic liver/renal disease
* Other concurrent severe and/or uncontrolled medical condition that could cause unacceptable safety risks/compromise compliance w protocol
* Treatment w any hematopoietic colony-stimulating factor ≤2wks prior to starting study drug. Erythropoietin is allowed
* Pts w history of CHF/arrhythmias who are receiving treatment w digoxin/verapamil, & treatment cannot be discontinued/switched to different drug prior to starting study drug
* Pts taking warfarin sodium
* Pts received treatment w PDGF/mTOR directed therapies
* Pts received chemo ≤ 4wks prior to starting study drug/have not recovered from side effects of such therapy
* Pts received immunotherapy ≤2 wks prior to starting study drug/have not recovered from side effects of such therapy
* Pts received investigational drugs ≤4 wks prior to starting study drug/have not recovered from side effects of such therapy
* Pts received XRT ≤4 wks prior to starting study drug/have not recovered from side effects of such therapy
* Pts undergone major non-CNS surgery ≤2 wks prior to starting study drug/pts have not recovered from side effects of such therapy
* Cardiac pacemaker, Ferromagnetic metal implants other than those approved as safe for use in MR scanners, Claustrophobia, Obesity
* Female pts are pregnant/breast feeding,/adults of reproductive potential not employing effective method of birth control. Barrier contraceptives must be used throughout trial in both sexes. Oral, implantable/injectable contraceptives may be affected by cytochrome P450 interactions, & are therefore not considered effective for study. Women of childbearing potential have negative serum pregnancy test 48hrs prior to administration of Gleevec, hydroxyurea and/or RAD001.
* Known diagnosis of HIV infection
* Pts w history of another primary malignancy that is currently clinically significant/currently requires active intervention
* Pts unwilling to/unable to comply w protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine MTD & DLT & Imatinib mesylate & RAD001 when combined w Hydroxyurea among pt w GBM | 6 months

SECONDARY OUTCOMES:
To further evaluate safety & tolerability & Imatinib mesylate in combo w RAD001 & Hydroxyurea | 6 months
To evaluate PK on Imatinib mesylate when administered w RAD001 among GBM pt who are on & not on EIAEDs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/